CLINICAL TRIAL: NCT04497935
Title: Comparative, Prospective and Randomized Study of Two Preparations for the Study of the Colon Through Colonoscopy
Brief Title: Comparison of Two Preparations for the Study of the Colon Through Colonoscopy
Status: Completed | Type: Observational
Sponsor: Unidade Local de Saúde do Alto Ave, EPE (Other)
Responsible Party: Principal Investigator, Cátia Vanessa Meixedo Arieira, Principal Investigator, Unidade Local de Saúde do Alto Ave, EPE
Other Study IDs: PLNV012018
Record Dates: First submitted 2020-07-28; First posted 2020-08-04 (Actual); Last update posted 2020-08-04 (Actual); Status verified 2020-07

CONDITIONS: Colon Cancer; Colon Polyp; Colon Adenoma; Colon Rectal Cancer
Keywords: Bowel preparation; Colonoscopy; Laxative
MeSH Terms: conditions — Colonic Neoplasms; Colonic Polyps | interventions — Polyethylene Glycols; MoviPrep

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (2):
- 1LPEG: Patients receiving 1LPEG who had a colonoscopy in the morning were advised to follow a day-before dosing regimen, where, at 7:00 pm the day before the colonoscopy, they prepared the Dose 1 sachet in 500 mL of water and consumed it over a period of 30 minutes, followed by 500 mL of clear liquids. The second dose was then taken at 11:00 pm by mixing the two Dose 2 sachets in a single glass of 500 mL of water and consuming them over 30 minutes, followed by 500 mL of clear liquids. If the colonoscopy was scheduled for the afternoon, the same dosing instructions were given, but the first dose was taken at 7:00 am on the day of the procedure, and the second dose began at 10:00 am.
  Interventions: Drug: PLENVU
- 2LPEG: Patients receiving 2LPEG who had a colonoscopy in the morning were asked to follow a similar day-before dosing regimen, where, at 7:00 pm the day before the colonoscopy, the first 1L dose was consumed over a 1-hour period, followed by the second dose at 11:00 pm. For 2LPEG patients with procedures in the afternoon, they took Dose 1 at 7:00 am and Dose 2 at 10:00 am. Any patient receiving 2LPEG was also told to consume 1L of clear liquids during the preparation procedure.
  Interventions: Drug: MoviPrep

INTERVENTIONS:
Drug: PLENVU — Bowel preparation for a colonoscopy
  Groups: 1LPEG
Drug: MoviPrep — Bowel preparation for a colonoscopy
  Groups: 2LPEG

SUMMARY:
Compare the quality of bowel preparation between two groups of patients, who will undergo two different preparations: 1. Moviprep + diet; 2. Plenvu + diet

DETAILED DESCRIPTION:
The quality of bowel preparation is essential for the success of a colonoscopy, reducing colonoscopy duration, and increasing the rate of cecal intubation and of polyp detection. There are several types of preparations available on the market and, irrespective of the choice, the split-dose regimen should be followed. A reduced volume preparation makes the process easier and more tolerable, increasing adhesion. Regarding the diet to be applied before the examination, there are no advantages to a liquid diet compared to a low fiber diet, and there is no evidence on the duration of the diet. In addition, a restrictive diet has an impact on satisfaction and also on adherence to treatment.

ELIGIBILITY:
Inclusion Criteria:

* All patients aged > 18 years and indicated for examination requiring bowel preparation

Exclusion Criteria:

* Pregnant or breastfeeding women
* Patients with gastroparesis or gastric obstruction.
* Patients with psychiatric disorders
* Severe renal impairment with CrCl <30mL/min
* Class III-IV Heart Failure
* Dependence / use of laxatives
* Chronic constipation (<3 stools/week).
* Uncontrolled hypertension (SBP >170mmHg or DBP >100mmHg)
* Intestinal Obstruction
* Colostomy from previous intestinal surgery
* Severe ascites
* Refusal of participation in the study
* Patients unable to understand or respond to the satisfaction survey

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients aged > 18 years and indicated for a colonoscopy requiring bowel preparation in the Gastroenterology Service of the Hospital of Senhora da Oliveira - Guimarães.
Sampling Method: Non-Probability Sample
Enrollment: 613 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2019-07-01 (Actual)

PRIMARY OUTCOMES:
Quality of bowel preparation between the two groups of patients | Patients were instructed to report any possible adverse events for up to 1 month after the procedure.
  The colonoscopist assessed each of the 3 colon segments on the BBPS and assigned each a score of 0 to 3. Successful overall bowel preparation is defined as a BBPS score of >6 with no individual segment scoring <2.

SECONDARY OUTCOMES:
Degree of satisfaction with the two bowel preparation | Patients were instructed to report any possible adverse events for up to 1 month after the procedure.
  The level of patient satisfaction with the 2 bowel preparation regimens was also assessed through a comparative analysis of the patient satisfaction questionnaire
Quality of bowel preparation in patients who had a morning or afternoon colonoscopy and those who received written, oral and additional telephone re-education on the day before the colonoscopy versus written and oral information only. | Patients were instructed to report any possible adverse events for up to 1 month after the procedure.
  The colonoscopist assessed each of the 3 colon segments on the BBPS and assigned each a score of 0 to 3. Successful overall bowel preparation is defined as a BBPS score of >6 with no individual segment scoring <2.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Senhora da Oliveira, Guimarães, Portugal